CLINICAL TRIAL: NCT03508440
Title: Intratympanic Steroid Injection for Treatment of Idiopathic Facial Nerve Paralysis
Brief Title: Intratympanic Steroid for Bell's Palsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Arnaldo L. Rivera, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007139
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Bell's Palsy; Facial Nerve Paresis
MeSH Terms: conditions — Bell Palsy | interventions — Injection, Intratympanic; Prednisone; Prednisolone

STUDY DESIGN:
Intervention Model Description: One arm will receive standard of care (SOC) in the form of high dose oral steroids for 10 days. The second arm will receive SOC plus 3 intratympanic steroid injections (space 7 days apart). Arm 3 is for patients who can not, for medical reasons, receive SOC; these patients will receive 3 intratympanic steroid injections (space 7 days apart).
Masking Description: There is no masking available as subject will know if they are receiving an intratympanic injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (Active Comparator): Oral steroids (prednisone or prednisolone) 60mg per day for 10 days or 60mg/day for 5 days followed by a 5 day taper
  Interventions: Drug: Prednisone
- SOC + injection (Experimental): Oral steroids as described above + intratympanic injection of dexamethasone (up to 1cc of 24mg/ml) - 3 injections over three weeks.
  Interventions: Procedure: Intratympanic injection; Drug: Prednisone
- Injection only (Other): Only Intratympanic injection of dexamethasone (up to 1cc of 24mg/ml) - 3 injections over three weeks
  Interventions: Procedure: Intratympanic injection

INTERVENTIONS:
Procedure: Intratympanic injection — Injection will be up to 1cc of dexamethasone 24mg/mL. The procedure will be performed at supine position under a microscope. Local anesthesia will be achieved with topical phenol. A myringotomy will be made in the tympanic membrane. A 1 mL syringe connected to a needle will be used to slowly inject between 0.2 cc and 1.0 cc of solution through the myringotomy, with the subject's head turned 45 degrees to the opposite side. The subject will be asked to maintain positioning for at least 30 minutes and refrain from swallowing. The dose administered will vary due to subject-specific factors.
  Arms: Injection only; SOC + injection
Drug: Prednisone — Oral Steroid
  Other Names: Prednisolone
  Arms: SOC + injection; Standard of Care

SUMMARY:
Facial nerve paralysis is due to inflammation around the facial nerve. Current treatment for facial nerve paralysis is a 10 day course of oral steroids (which will reduce the inflammation), with electrodiagnostic testing. There have been limited studies on the use of intratympanic steroid injection, in addition to oral steroid, in the recovery of facial nerve paralysis. There are indications that the use of intratympanic injections, in addition to the oral steroids, will speed up the recovery rate of the facial nerve paralysis, as well as improve the complete recovery of the facial nerve paralysis. This study will randomize patients with facial nerve paralysis into two groups: 1) oral steroid only and 2) oral steroid plus a 3 intratympanic steroid injections spaced out over three weeks. There are a subset of patients that are unable to take oral steroids for medical reasons (such as diabetes); these patients will be placed into a third group and only receive 3 intratympanic steroid injections space out over three weeks. Subjects that are to receive the intratympanic injection will receive pre- and post-hearing exams as part of their standard of care. Patients will be evaluated via videorecording by two blinded investigators as well as in person evaluations by the unblinded treating physician.

Subjects will be followed until complete facial nerve paralysis recovery or one year post-treatment, whichever comes first.

DETAILED DESCRIPTION:
Facial nerve paralysis is due to inflammation surrounding the facial nerve. Current clinical practice guidelines for treatment of facial nerve paralysis recommend a 10 day course of oral steroids +/- oral acyclovir. Treatment should begin within 72 hours of symptom onset. In patients with complete facial paralysis, electrodiagnostic testing should be offered to the patient (1-2). In patients with 90% degeneration on electroneuronography (ENoG) testing, facial nerve decompression may be considered but is not a current recommendation.

In 1973, Bryant reported on ten cases where intratympanic steroid injection was used for the treatment of Bell's palsy (3). All but one of these patients had complete recovery of their facial nerve function. The remaining patient had 75% recovery. None of these patients suffered complications from the injections. The next study published on intratympanic steroid injection for Bell's palsy was not published until 2014 (4). It was a randomized control trial that divided patients into standard treatment (oral steroids and acyclovir) versus standard treatment with intratympanic steroid injection. There was not a statistically significant difference between the complete recovery rate of the control group and of the intratympanic steroid group; however, the time to recovery was significantly shorter in the intratympanic steroid injection group as compared to the control group. Limitations of this study include small sample size and high attrition rate.

There have not been any other studies published in the literature looking at improving facial nerve recovery in idiopathic facial nerve paralysis with the use of intratympanic steroid injections.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language
* Acute unilateral facial palsy without skin lesions which developed within a 72-hour period and is present for 21 days or less.
* Moderate to severe facial palsy [House-Brackmann grade IV or greater]

Exclusion Criteria:

* Another cause of facial nerve paralysis that is not idiopathic
* Otologic disease including otitis media, temporal bone fracture, a previous history of facial nerve palsy in either side, history of otologic surgery, and suspected Ramsay Hunt syndrome.
* Systemic disease including history of tuberculosis, history of head and neck cancer, other neurological disorders, recent use of ototoxic medications, liver or renal dysfunction, and other illnesses that would contraindicate the use of high-dose steroid therapy.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo Rivera, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable...we do not plan to share individual participant data with other researchers so that we can maintain the privacy of our participants.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | SOC + Injection | Injection Only
Started | 1 | 9 | 0
Completed | 1 | 9 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Injection only was for participants who could not, for medical reasons, receive the SOC treatment. We did not have any patients that met that criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | SOC + Injection | Injection Only | Total
Number analyzed (Participants) | 1 | 9 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (0) | 52.90 (13.836) |  | 52.90 (13.836)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 |  | 3
  Male | 0 | 7 |  | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 9 |  | 10
House Brackman Score at Diagnosis [Mean (Standard Deviation); unit: units on a scale] — Grading system that measures the degree of facial nerve damage in a patient with facial palsy.
  Minimum score is 1: normal function; no facial palsy Maximum score is 6: total paralysis; no movement
  units on a scale | 5 (0) | 5.11 (0.928) |  | 5.10 (0.876)

OUTCOME MEASURES:

1. Primary Outcome: Facial Nerve Recovery
Description: Time (in days) from the diagnosis or start of treatment to complete recovery of paralysis, defined as house brackman score of 1
Time Frame: Up to 365 days
Population: Adults over the age of 18 that presented with Bell's palsy and a House Brackman score of 4 or greater
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard of Care | SOC + Injection | Injection Only
Number analyzed (Participants) | 1 | 9 | 0
Days | 7 (0) | 81.56 (47.671) |

ADVERSE EVENTS:
Time Frame: For each patient, AE's were collected from the time of informed consent until complete facial nerve paralysis recovery or one year post-treatment, whichever comes first
Description: We used the definition of AE as defined by Clinicaltrials.gov
Arm/Group | Standard of Care | SOC + Injection | Injection Only
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/9 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03508440/Prot_SAP_001.pdf